CLINICAL TRIAL: NCT00409305
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Examine the Effect of Betahistine on Body Weight in Obese Subjects
Brief Title: The Effect of Betahistine on Body Weight in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OBEcure Ltd. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BET201
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2007-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Betahistine; Nutrition Assessment

INTERVENTIONS:
Drug: Betahistine
Behavioral: Dietary counseling

SUMMARY:
The purpose of this study is to examine the effect that betahistine has on body weight in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Male or female subjects 18 to 65 years of age;
* Is obese with a BMI greater than or equal to 30 kg/m2 to less than or equal to 40 kg/m2;
* Has been obese for at least 1 year prior to screening; and
* If female, is nonlactating, has a negative urine pregnancy test result, and does not plan on becoming pregnant during the study, or not of childbearing potential (hysterectomy or tubal ligation at least 6 months prior to randomization or post-menopausal for 1 year); if of childbearing potential (including peri-menopausal women who have had a menstrual period within 1 year) must practice or be willing to continue to practice appropriate birth control (such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire study duration.

Exclusion Criteria:

* Has obesity of known endocrine origin (e.g., Cushing's disease, Addison's disease, hypothalamic tumor);
* Has a medical history (e.g., morbid childhood obesity) and/or physical characteristics (e.g., polydactyly) suggestive of genetic obesity (e.g., ob/ob genotype) or syndromatic obesity (e.g., Prader-Willi syndrome, Bardet Biedl syndrome);
* Previous surgical procedures for weight loss;
* Has had liposuction within 1 year before screening or is planning to have liposuction during the study;
* History of bulimia or evidence of laxative abuse;
* Has had a body weight loss of >4 kg in the 90 days prior to screening;
* Has taken drugs capable of influencing body weight 30 days prior to screening;
* Has recently started or plans on starting a smoking cessation program;
* Has had a major change in daily physical activity (e.g., initiation of an exercise program) or started a weight loss program within 90 days prior to screening;
* Is unwilling or unable to participate in a dietary program as part of the study;
* Is <80% compliant with study medication in the single-blind placebo run-in period;
* Has a clinically significant history or presence of any of the following conditions:
* Active or past history of cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities;
* Liver disease (irrespective of transaminase concentrations);
* Pheochromocytoma;
* Porphyria;
* Type 1 diabetes mellitus;
* Type 2 diabetes mellitus on treatment other than metformin monotherapy and/or diet with HbA1c less than or equal to 8%;
* Severe type 2 diabetes with history of ketoacidosis or diabetic ulcers, or presence of retinopathy, neuropathy, or nephropathy;
* Renal insufficiency defined as a serum creatinine greater than or equal to 1.5 mg/dL (133 µmol/L) at screening;
* Malignant disease within 5 years of screening;
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x ULN;
* Thyroid-stimulating hormone (TSH) outside of the normal range;
* Plans on having any surgery (elective or otherwise) during the course of the study;
* Has uncontrolled hypertension (sitting blood pressure >160/95 mmHg at screening or randomization), uncontrolled hyperlipidemia (triglycerides [TG] greater than or equal to 400 mg/dL or low-density lipoprotein cholesterol [LDL-C] >160 mg/dL), or uncontrolled diabetes (HbA1c >8%);
* History of asthma;
* History of peptic ulcers;
* History of HIV;
* History of undiagnosed allergy, severe allergy, or drug allergy, including history of anaphylaxis, angioedema, bronchospasm, or urticaria;
* Has clinical laboratory test values (chemistry, hematology, or urinalysis) judged to be clinically significant by the investigator;
* Has a physical examination or electrocardiogram (ECG) with significant abnormalities, as judged by the investigator;
* Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion could cause the subject to be noncompliant with study procedures;
* Has hypersensitivity to betahistine;
* Has psychiatric or neurological disorders requiring chronic medications (e.g., antidepressants), subjects are to be unlikely to have a major depressive episode (score of lees than or equal to 8) on The Harvard Department of Psychiatry and National Depression Screening Day Scale (THE HANDS) (See Appendix E);
* Chronic or as needed use of antihistamines;
* Has not been on a stable treatment regimen with any of the following medications for a minimum of 90 days prior to screening:
* Hormone replacement therapy;
* Oral contraceptives;
* Antihypertensive agents;
* Metformin;
* Lipid-lowering agents; or
* Thyroid replacement therapy;
* Has been treated over the past 60 days, is currently treated, or is expected to require or undergo treatment with any of the following excluded medications;
* All prescription or over-the-counter agents taken for the purpose of weight reduction, including (but not limited to) the following anti obesity agents:
* Prescription drugs such as orlistat, sibutramine, and phentermine; or
* Over-the-counter antiobesity agents (e.g., herbal supplements or other alternative remedies such as Cortislim, Dexatrim, Acutrim);
* Psychotropic/neurological agents including the following:
* Antipsychotic agents (e.g., olanzapine, clozapine, risperidol, lithium, etc.).
* Antiepileptic agents (e.g., Topamax®, Zonegran®, valproate, carbamazepine); or
* Antidepressant agents including the following: monoamine oxidase inhibitors, bupropion (Wellbutrin®, Zyban®), tricyclic antidepressants, and tetracyclic antidepressants; and selective serotonin reuptake inhibitors (e.g., Prozac®, Paxil®, Zoloft®, etc.);
* Systemic steroids administered by oral, intravenous, or intramuscular route;
* Drugs that directly affect gastrointestinal motility (e.g., Reglan® and Propulsid®, and chronic [taken for more than 10 days within a 6-month period] macrolide antibiotics such as erythromycin and newer derivatives);
* Calcitonin (e.g., Miacalcin®);
* Insulin;
* Exenatide (Byetta);
* Sulfonylureas (e.g., Diamicron, Amaryl, Glucotrol, Micronase); or Meglitinides (e.g., Starlix, Prandin)
* Has received any investigational drug within 90 days of screening;
* Receipt of any investigational treatment (drug or device) within 90 days prior to screening;
* Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site; or
* Is employed by OBEcure Ltd.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2007-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To examine the effect of betahistine on body weight in obese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ahmann, MD, Principal Investigator — Covance CRU, Inc; Louis Aronne, MD, Principal Investigator — Comprehensive Weight Control Program; Harold Bays, MD, Principal Investigator — L-Marc Research Center; Norman Fishman, MD, Principal Investigator — Diabetes & Endocrinology Specialists; Ken Fujioka, MD, Principal Investigator — Scripps Clinic, Nutrition Metabolic Research; Jeffrey Geohas, MD, Study Director — Radiant Research, Inc; Frank Greenway, MD, Principal Investigator — Pennington Biodmedical Research Center; Dean Kereiakes, MD, Principal Investigator — Lindner Clinical Trial Center; Diane Krieger, MD, Principal Investigator — Miami Research Associates, Nutrition Division; Robert Kushner, MD, Principal Investigator — NCCR; Thomas Moretto, MD, Principal Investigator — American Health Network; Monica Pierson, MD, Principal Investigator — Radiant Research; Sherwyn Schwartz, MD, Principal Investigator — Diabetes & Glandular Disease Research Associates; Diane Smith, MD, Principal Investigator — CSRA Partners in Health; Philip Toth, MD, Principal Investigator — Midwest Institute for Clinical Research; Mervyn Weerasinghe, MD, Principal Investigator — Rochester Clinical Research; Richard Weinstein, MD, Principal Investigator — Diablo Clinical Research; Lisa Wright, MD, Principal Investigator — Cahaba Research, Inc; James Zavoral, MD, Principal Investigator — Radiant Research, Inc.; Nir Barak, MD, Study Director — OBEcure Ltd.; Yaffa Beck, PhD, Study Chair — OBEcure Ltd.; Ami Eyal, MD, Study Chair — OBEcure Ltd.
Locations (19):
- United States (19):
  - Cahaba Research, Inc., Birmingham, Alabama
  - Scripps Clinic, Nutrition Metabolic Research, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Miami Research Associates, Inc., Nutrition Division, Miami, Florida
  - CSRA Partners in Health, Inc., Augusta, Georgia
  - Radiant Research, Inc., Chicago, Illinois
  - NCCR, Chicago, Illinois
  - American Health Network, Indianapolis, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Radiant Research, Inc., Overland Park, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Radiant Research, Inc., Edina, Minnesota
  - Diabetes & Endocrinology Specialists, Chesterfield, Missouri
  - Comprehensive Weight Control Program, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Covance CRU, Inc., Portland, Oregon
  - Diabetes & Glandular Disease Research Associates, Inc., San Antonio, Texas